CLINICAL TRIAL: NCT00874289
Title: Utility of NGAL in Predicting Renal Impairment, Further Decompensation & Rehospitalization in Acutely Decompensated & Chronic Heart Failure Patients
Brief Title: Utility of Neutrophil Gelatinase-associated Lipocalin (NGAL) in Predicting Renal Impairment, Further Decompensation and Rehospitalization in Acutely Decompensated and Chronic Heart Failure Patients
Acronym: ANGLE-HF
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Collaborators: Abbott RDx Cardiometabolic (Other)
Responsible Party: Principal Investigator, Henry Krum, Prof Henry Krum, The Alfred
Other Study IDs: CP-01/08
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Heart Failure
Keywords: NGAL; Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples are being collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute heart failure patients
  Interventions: Other: NGAL kit
- Chronic heart failure patients
  Interventions: Other: NGAL kit

INTERVENTIONS:
Other: NGAL kit — Kit to test NGAL levels in heart failure patients

SUMMARY:
Acute decompensated heart failure (ADHF) is the leading cause of admission to hospital in the US, and is associated with high mortality, morbidity, and major cost to the health care system. Much of this cost relates to prolonged hospitalizations from acute deterioration in kidney function (AKI), which in turn is associated with further cardiovascular events such as recurrent ADHF. Strategies for early detection minimization and prevention of AKI would therefore be of tremendous benefit to both the patient and the health care system.

A common reason for hospitalization in ADHF is that of altered volume status and renal impairment. Also, many patients with ADHF have underlying hypertension and/or a recent acute coronary syndrome. Hypertension, diabetes and chronic kidney disease (CKD) are independent risk factors for cardiovascular disease, and diabetes is the leading cause of CKD. Therefore, patients presenting with ADHF are at high risk for CV events, more so if they develop AKI. Therefore, strategies to detect changes in renal status early may allow for more rapid intervention with appropriate drug and other therapies to attenuate AKI and subsequent complications, which may in turn result in prevention of early readmissions with HF.

Most ADHF patients have underlying chronic heart failure (CHF). CHF is a major cost to the health care system. About two thirds of this cost relates to hospitalization for acute deterioration in heart failure (HF). Strategies to minimize or prevent HF hospitalization therefore are of tremendous benefit to both the patient and the health care system.

The most frequent reason for hospitalization in a CHF patient is that of altered volume status and renal impairment. Therefore, as with ADHF, strategies for early detection of changes in renal status may allow for intervention with appropriate drug and other therapies to attenuate, or even prevent, the need for the patient to return to hospital.

Many approaches have been studied in relation to this concept. Deterioration in renal function is a harbinger of a need for hospitalization, and indeed a predictor of medium term mortality. However, current measures of renal function are relatively crude with a considerable lag between an insult to the kidney and its translation to a measurable deterioration in renal function reflected by worsening serum creatinine. Thus, diagnostic tests that evaluate renal injury which are modulated early in the time course of this process may have considerable utility not only in the ADHF setting but also in predicting decompensation in the CHF setting.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females
2. Age >18years
3. Confirmed written informed consent
4. Acute decompensated heart failure cohort defined as:

   * Objective evidence of heart failure (of any cause/etiology) demonstrated by typical symptoms/signs combined with an imaging modality (see appendix for criteria)
   * Requirement for intravenous diuretic whilst either an inpatient or in an emergency room setting with intravenous diuretics, vasodilators or inotropes
   * No ejection fraction cut-off will be required, ie both systolic and diastolic heart failure patients can be enrolled
5. Chronic Heart Failure cohort defined as:

   * Echocardiographic evidence of systolic or diastolic heart failure (see appendix for criteria)
   * CHF patients in Class III and class IV NYHA symptoms who have had a minimum of one acute decompensated episode in the previous six months
   * Evidence of impaired renal function (eGFR <60 ml/min)

Exclusion Criteria:

1. Patients with a history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study
2. Not meeting entry criteria for ADAF (as above)
3. At the discretion of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute and chronic heart failure
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2008-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To assess the utility of NGAL in predicting death, rehospitalisation or deterioration of renal function (increase in creatinine of >0.3 mmol/L) at 12 months | 12 months

SECONDARY OUTCOMES:
To assess the utility of NGAL in predicting subsequent HF rehospitalisation and predicting clinical deterioration, ie worsening symptoms and/or signs (based on NYHA class) at 30, 90 days (ADHF patients), 6 months and 12 months (CHF patients) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, MBBS FRACP PhD, Principal Investigator — Monash University / Alfred Hospital
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia